CLINICAL TRIAL: NCT06837883
Title: The Impact of Through-and-through Guidewire on the Outcome of Percutaneous Nephrolithotomy (PCNL) in Complex Renal Stones: a Randomized Controlled Study
Brief Title: The Impact of Through-and-through Guidewire on Percutaneous Nephrolithotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Osama Mahmoud, Dr., South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URO016/4/624
Record Dates: First submitted 2025-02-17; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Nephrolithotomy, Percutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group using through and through guiedwire (Experimental): In the study group, a modification was carried out to have through-and-through guidewire. The procedure begins with the retrograde insertion of 2 guidewires, followed by the insertion of the ureteral catheter via one of the two guidewires. Percutaneous access is performed as usual. Using rigid nephroscopy or ureteroscopy, the guidewire was pulled antegrade through the access sheath to create a through-and-through guidewire. If it is difficult to access the guidewire, stone fragmentation is initiated and the guidewire is pulled out during the procedure. Otherwise, the procedure is performed as described above. If a post-operative DJ stent is required, we use the through-and-through guidewire directly for insertion.
  Interventions: Procedure: Percutaneous nephrolithotomy through and through guiedwire
- Standard percutaneous nephrolithotomy (Active Comparator): In the control group, the procedure began with the insertion of a ureteral catheter in the lithotomy position, followed by percutaneous renal puncture in the prone position under fluoroscopic guidance. A nitinol-PTFE hybrid guidewire was inserted through the needle and initially guided towards the ureter, with difficulty entering the ureter, tract dilation was performed according to the guidewire position. Tracts were dilated to 28Fr using Alken's dilators and a 24-F rigid nephroscopy (Karl Storz, Germany) was used. Stones were disintegrated with pneumatic lithotripsy (Swiss Lithoclast Master, EMS, Nyon, Switzerland) and fragments were extracted with forceps or stone basket. For inacessible stones, a flexible cystoscopy (Karl Storz, Flex X2, GmbH) and laser disintegration was used (holmium:YAG laser: Versa Pulse PowerSuit 20 W; Lumenis Inc., Dreieich-Dreieichenhain, Germany).
  Interventions: Procedure: Standard percutaneous nephrolithotomy

INTERVENTIONS:
Procedure: Percutaneous nephrolithotomy through and through guiedwire — In the study group, a modification in percutaneous nephrolithotomy was carried out to have through-and-through guidewire.
  Arms: Study group using through and through guiedwire
Procedure: Standard percutaneous nephrolithotomy — Standard percutaneous nephrolithotomy without using through and through guide wire
  Arms: Standard percutaneous nephrolithotomy

SUMMARY:
The aim to the study is to investigate the impact of combined retrograde and antegrade insertion of a through-and-through guidewire during percutaneous nephrolithotomy (PCNL). Adult patients with complex renal stones (Guy's stone score III, IV) were ranomized between standard PCNL (control group) and PCNL with comibined retrograde and antegrade inserted through-and-through guidewire (study group). This modification initially involves the retrograde insertion of an additional guidewire beside the ureteral catheter. After percutaneous puncture and dilation of the tract, the guidewire is pulled antegrade through the renal access, using either ureteroscopy or nephroscopy to secure the tract throughout the procedure.The primary outcome is to compare the initial stone free rate (SFR) between both groups. The secondary outcome is to compare both groups as regard operative time, fluorscopy time, number of tracts, haemoglobin drop, blood transfusion and major complications accoridng to Clavien-Dindo (CD) system. Success is defined as presence of insignificant residual less than 4 mm.

DETAILED DESCRIPTION:
Intervention All patients underwent PCNL under general anesthesia. In the control group, the procedure began with the insertion of a ureteral catheter in the lithotomy position, followed by percutaneous renal puncture in the prone position under fluoroscopic guidance. A nitinol-PTFE hybrid guidewire was inserted through the needle and initially guided towards the ureter, with difficulty entering the ureter, tract dilation was performed according to the guidewire position. Tracts were dilated to 28Fr using Alken's dilators and a 24-F rigid nephroscopy (Karl Storz, Germany) was used. Stones were disintegrated with pneumatic lithotripsy (Swiss Lithoclast Master, EMS, Nyon, Switzerland) and fragments were extracted with forceps or stone basket. For inacessible stones, a flexible cystoscopy (Karl Storz, Flex X2, GmbH) and laser disintegration was used (holmium:YAG laser: Versa Pulse PowerSuit 20 W; Lumenis Inc., Dreieich-Dreieichenhain, Germany). If it was difficult to reach the stones with the flexible nephroscopy, additional tracts were used. At the end of the procedure, an 18-20 F nephrostomy tube was left in each tract for 24-48 hours. In some cases where the pelvic-caecal system is injured or multiple significant residuals are present, an antegrade DJ stent is placed by withdrawing the ureteral catheter and inserting a guidewire up to the bladder to then replace the ureteral catheter with a DJ stent.

In the study group, a modification was carried out to have through-and-through guidewire. The procedure begins with the retrograde insertion of 2 guidewires, followed by the insertion of the ureteral catheter via one of the two guidewires. Percutaneous access is performed as usual. Using rigid nephroscopy or ureteroscopy, the guidewire was pulled antegrade through the access sheath to create a through-and-through guidewire. If it is difficult to access the guidewire, stone fragmentation is initiated and the guidewire is pulled out during the procedure. Otherwise, the procedure is performed as described above. If a post-operative DJ stent is required, we use the through-and-through guidewire directly for insertion.

Surgical data such as operative time starting by the percutaneous puncture, total fluoroscopy time, number of tracts and complications are recorded. On the on the 1st postoperative day, both US and plain X-rays were used to assess stone free rate for the radiopaque stones, while for radiolucent stone NCCT is used.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients without contraindications for PCNL with Guy's stone score III-IV were randomized to either standard PCNL (control group) or PCNL with retrograde and antegrade inserted through-and-through guidewire (study group)

Exclusion Criteria:

* solitary or solitary functioning kidney, renal congenital anomlalies, and urinary diversion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Stone free rate (SFR) between both groups | within one week postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Osama Mahmoud, Dr., Principal Investigator — South Valley University
Locations (1):
- Qena Faculty of Medicine, Qina, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All the the individual data collected during the trial will be available, after deidentification
Supporting Information: Study Protocol
Time Frame: After publication without time limit
Access Criteria: Anyone who wishes to access the data